CLINICAL TRIAL: NCT06469112
Title: The Effect of Vibration on Pain During Subcutaneous Heparin Injection: A Randomized Controlled Study
Brief Title: The Effect of Vibration on Pain During Subcutaneous Heparin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Associate Professor, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-28/1
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-01

CONDITIONS: Pain; Asthma; Pulmonary Disease; Chest Disorder
Keywords: Subcutaneous heparin injection; pain; non-pharmacological method; vibration
MeSH Terms: conditions — Pain; Asthma; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Vibration Application Group (Experimental): With individuals in this group, device will be used to provide vibration. This device, designed as a combination of cold application and local vibration to reduce pain experienced during invasive procedures, is frequently chosen for all age groups. There is a motor in the body which provides vibration. The device also has ice wings behind the body, which are used to provide cold, but these will not used in this research.
  The device, at room temperature, was placed by the researcher 5 cm proximal to the injection site before the injection will performed. For one minute before the injection, a slight non-discomforting vibration will make, and this will be continue while the injection was given. In this study, only the body of the device will be used to provide vibration.
  Interventions: Device: Vibration
- Placebo: Intervention Control Group (Placebo Comparator): The device was used with participants in this group. The device, at room temperature, was placed by the researcher 5 cm proximal to the injection site before the injection was performed. With participants in this group, the device was placed on the procedure site, but no vibration was made. The device was held on the participants for one minute before the injection and throughout the procedure, with the vibration switched off.
  Interventions: Other: Placebo
- Control: Nonintervention Group (No Intervention): No intervention was performed before or during the procedure with the participants in the control group, and the standard subcutaneous heparin injection procedure was carried out.

INTERVENTIONS:
Device: Vibration — The device was used to provide vibration with the participants in this group. This device, designed as a combination of cold application and local vibration to reduce pain experienced during invasive procedures, is frequently chosen for all age groups.
  Arms: Experimental: Vibration Application Group
Other: Placebo — The device was used with participants in this group. The device, at room temperature, was placed by the researcher 5cm proximal to the injection site before the injection was performed. With participants in this group, the device was placed on the procedure site, but no vibration was made. The device was held on the participants for one minute before the injection and throughout the procedure, with the vibration switched off.
  Arms: Placebo: Intervention Control Group

SUMMARY:
Aim: The aim of this research will to examine the effect of the local vibration technique applied to the injection site during subcutaneous low molecular weight heparin (LMWH) injection.

Methods: The patients will randomly assigned to an experimental (vibration) group , a placebo control group, and a nonintervention control group. Participants in the experimental group will give slight vibration to the injection site before the injection will administered; for participants in the placebo group, the device will placed on the injection site but with the vibration button kept switched off, while for the nonintervention control group, routine subcutaneous low molecular weight heparin injection will administered. The level of pain felt by the participants during the administration of the injection will assess with a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* being over the age of 18
* having a doctor's prescription for subcutaneousheparin 0.6 mL treatment with a ready-to-use syringe and not yet having begun treatment
* having no coagulation disorder
* having no disorder which could affect pain perception,
* having no incision, lipodystrophy or finding of infection at the injection site,
* having no communication problem, and voluntarily agreeing to participate in the research

Exclusion Criteria:

* being under the age of 18
* having diabetes mellitus
* peripheral vascular disease, etc. which could affect the perception of pain
* not being conscious, refusing to participate in the research or opting to leave the study at any point.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
pain intensity in mm | 6 months
  A 10-cm vertical VAS will used to evaluate the severity of pain felt by the individuals during the procedure. One end indicated lack of pain and the other the most severe pain possible.

SECONDARY OUTCOMES:
weight | 6 months
  weight in kilograms
height | 6 months
  height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided